CLINICAL TRIAL: NCT05844423
Title: Randomized, Observer-Blind, Active-Controlled, Dose-Finding Study to Evaluate the Safety, Tolerability, and Immunogenicity of 24-Valent PCV (VAX-24) in Infants Given 4 Doses at 2, 4, 6, and 12-15 Months of Age With Pediatric Vaccines
Brief Title: Safety, Tolerability, and Immunogenicity of a 24-Valent Pneumococcal Conjugate Vaccine (VAX-24) in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vaxcyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAX24-112
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pneumococcal Vaccines
Keywords: 24 valent PCV; Pneumonia; Pneumococcal Infection
MeSH Terms: conditions — Pneumonia; Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VAX-24 Low (Experimental): Participants will receive 4 doses of VAX-24 administered as an intramuscular injection at 2, 4, 6, and 12-15 months of age at one of three dose levels.
  Interventions: Biological: 0.5 ml dose of 1.1 mcg VAX-24
- VAX-24 Mid (Experimental): Participants will receive 4 doses of VAX-24 administered as an intramuscular injection at 2, 4, 6, and 12-15 months of age at one of three dose levels.
  Interventions: Biological: 0.5 ml dose of 2.2 mcg VAX-24
- VAX-24 Mixed (Experimental): Participants will receive 4 doses of VAX-24 administered as an intramuscular injection at 2, 4, 6, and 12-15 months of age at one of three dose levels.
  Interventions: Biological: 0.5 ml dose of 2.2/4.4 mcg VAX-24
- PCV20 (Active Comparator): Participants will receive 4 doses of PCV20 administered as an intramuscular injection of the standard dose at 2, 4, 6, and 12-15 months of age.
  Interventions: Biological: 0.5 ml dose of PCV20

INTERVENTIONS:
Biological: 0.5 ml dose of 1.1 mcg VAX-24 — 24 valent pneumococcal conjugate vaccine
  Arms: VAX-24 Low
Biological: 0.5 ml dose of PCV20 — 20 valent pneumococcal conjugate vaccine
  Arms: PCV20
Biological: 0.5 ml dose of 2.2 mcg VAX-24 — 24 valent pneumococcal conjugate vaccine
  Arms: VAX-24 Mid
Biological: 0.5 ml dose of 2.2/4.4 mcg VAX-24 — 24 valent pneumococcal conjugate vaccine
  Arms: VAX-24 Mixed

SUMMARY:
The objective of the study is to evaluate the safety and tolerability of 4 injections of VAX-24 (at 3 dose levels) compared to PCV15 in infants at 2, 4, 6, and 12-15 months of age, in addition to receiving routine US concomitant vaccines. Stage 1 of the study will comprise 3 dose ascending cohorts. Stage 2 of the study will enroll the remainder of the sample size.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female infant ≥42 days to ≤89 days (inclusive).
2. Full-term infant at least 37 weeks gestational age at birth.
3. Afebrile for ≥72 hours with a rectal temperature <38.0°C (<100.4°F) or axillary temperature <37.8°C (<100.0°F) before receipt of study vaccine.*
4. Able to attend all scheduled visits and comply with the study procedures.
5. Subject's parent/legal guardian is able to read and understands the study procedures, alternate treatments, risks and benefits, and provides written informed consent.
6. Subject's parent/legal guardian is able to fill out an ediary of solicited AE and take daily axillary temperature and measurements of local injection site reactions for the 7 days after each study vaccination.
7. Subject's parent/legal guardian has an e-mail address and access to a computer or smartphone with internet to complete the ediary.

Exclusion Criteria:

1. History of invasive pneumococcal disease (positive blood culture, positive cerebrospinal fluid culture, or other sterile site) or known history of other culture positive pneumococcal disease.
2. Previous receipt of a licensed or investigational vaccine (excluding 1 dose hepatitis B vaccine).
3. Known hypersensitivity to any vaccine.
4. Known or suspected impairment of immunological function (e.g., asplenia, HIV, primary immunodeficiency).
5. Use of any immunosuppressive therapy (Note: topical and inhaled/nebulized steroids are permitted).
6. History of failure to thrive.
7. Subject has a coagulation disorder contraindicating IM vaccination.
8. Subject or his/her mother have documented hepatitis B surface antigen-positive.
9. Has a known neurologic or cognitive behavioral disorder.
10. Has a known clinically significant congenital malformation or serious chronic disorder.
11. Receipt of a blood transfusion or blood products, including immunoglobulins.
12. Receipt of any investigational study product since birth, currently participating in another interventional investigational study, or having plans to receive another investigational product(s) while on study.
13. Any infant who cannot be adequately followed for safety according to the protocol plan.
14. Any other reason that in the opinion of the investigator may interfere with the evaluation required by the study.

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 802 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with any solicited local injection site Adverse Events (AE) within 7 days after each vaccination | 7 days after each vaccination
  Solicited local reactions include erythema, edema, and tenderness at the injection site
Percentage of participants with any solicited systemic AE within 7 days after each vaccination | 7 days after each vaccination
  Solicited systemic reactions include fever, irritability, decreased appetite, decreased sleep, and increased sleep
Percentage of participants with any related Serious Adverse Events (SAE) within 6 months after last vaccination | 6 months after last vaccination
  Percentage of participants with related SAE

SECONDARY OUTCOMES:
Percentage of subjects with any unsolicited AE within 1 month after each vaccination | 1 month after each vaccination
  Percentage of subjects with any unsolicited AE
Percentage of subjects with any unsolicited AE from Dose 1 through 1 month post-Dose 3 | First vaccination (Dose 1) through 1 month after third vaccination (Dose 3)
  Percentage of subjects with any unsolicited AE between first and 3rd vaccination in the primary series
Percentage of subjects with any AE resulting in discontinuation of study within 6 months after last vaccination | 6 months after last vaccination
  Percentage of subjects with any AE resulting in discontinuation of study
Percentage of subjects with any new onset of chronic illness (NOCI) within 6 months after last vaccination | 6 months after last vaccination
  Percentage of subjects with any NOCI
Percentage of subjects with any medically attended adverse events (MAAE) within 6 months after last vaccination | 6 months after last vaccination
  Percentage of subjects with any MAAE
Percentage of subjects with any SAE within 6 months after last vaccination | 6 months after last vaccination
  Percentage of subjects with any SAE
Percentage of subjects achieving an anti-pneumococcal Immunoglobulin G (IgG) antibody concentration ≥0.35 mcg/mL 1 month after Dose 3 | 1 month after Dose 3
  Percentage of subjects achieving an anti-pneumococcal IgG antibody concentration ≥0.35 mcg/mL
Percentage of subjects achieving an anti-pneumococcal IgG antibody concentration ≥0.35 mcg/mL 1 month after Dose 4 | 1 month after Dose 4
  Percentage of subjects achieving an anti-pneumococcal IgG antibody concentration ≥0.35 mcg/mL
IgG antibody Geometric Mean Concentration (GMC) 1 month after Dose 3 | 1 month after Dose 3
  Antibody geometric mean concentrations as measured by IgG for the 24 pneumococcal serotypes in VAX-24
IgG antibody GMC 1 month after Dose 4 | 1 month after Dose 4
  Antibody geometric mean concentrations as measured by IgG for the 24 pneumococcal serotypes in VAX-24
Opsonophagocytic activity (OPA) Geometric Mean Titer (GMT) 1 month after Dose 3 | 1 month after Dose 3
  Antibody geometric mean titers s as measured by OPA for the 24 pneumococcal serotypes in VAX-24
OPA GMT 1 month after Dose 4 | 1 month after Dose 4
  Antibody geometric mean titers s as measured by OPA for the 24 pneumococcal serotypes in VAX-24
IgG Geometric Mean Fold Ratio (GMFR) before Dose 4 to 1 month after Dose 4 | Pre-Dose 4 to 1 month after Dose 4
  Antibody geometric mean fold ratio as measured by IgG for the 24 pneumococcal serotypes in VAX-24
OPA GMFR before Dose 4 to 1 month after Dose 4 | Pre-Dose 4 to 1 month after Dose 4
  Antibody geometric mean fold rise as measured by OPA for the 24 pneumococcal serotypes in VAX-24
Percentage of subjects achieving at least a 4-fold increase in IgG from pre-Dose 4 to 1 month post Dose 4 | Pre-Dose 4 to 1 month after Dose 4
  Geometric mean concentration with a at least a 4-fold increase in IgG antibodies for the 24 pneumococcal serotypes in VAX-24
Percentage of subjects achieving at least a 4-fold increase in OPA titers from pre-Dose 4 to 1 month post Dose 4 | Pre-Dose 4 to 1 month after Dose 4
  Geometric mean titer with a at least a 4-fold increase in OPA titers for the 24 pneumococcal serotypes in VAX-24

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Madera Family Medical Group, Madera, California
  - Jedidiah Clinical Research, Tampa, Florida
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - ACC Pediatric Research, Haughton, Louisiana
  - Meridian Clinical Research, Hastings, Nebraska
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Ohio Pediatric Research Assn., Dayton, Ohio
  - UPMC Bass Wolfson Cranberry, Cranberry Township, Pennsylvania
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - UPMC Children's Community Pediatrics South Hills-Jefferson Hills, Jefferson Hills, Pennsylvania
  - UPMC Primary Care Center Oakland, Pittsburgh, Pennsylvania
  - UPMC Children's Community Pediatrics Bass Wolfson-Squirrel Hill, Pittsburgh, Pennsylvania
  - UPMC Children's Community Pediatrics-Castle Shannon, Pittsburgh, Pennsylvania
  - Palmetto Pediatrics, PA, North Charleston, South Carolina
  - Tribe Clinical Research at Parkside Pediatrics, Simpsonville, South Carolina
  - Coastal Pediatric Research, Summerville, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Ventavia Research Group, Burleson, Texas
  - Ventavia, Houston, Texas
  - Kool Kids Pediatrics, Houston, Texas
  - Pediatric Associates, Houston, Texas
  - Pediatric Center, Richmond, Texas
  - Alliance for Multispecialty Research, Layton, Utah
  - Alliance for Multispecialty Research, Murray, Utah
  - Alliance for Multispecialty Research, Provo, Utah
  - Alliance for Multispecialty Research, Roy, Utah
  - Alliance for Multispecialty Research, Syracuse, Utah
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Vaxcyte is committed to providing access to anonymized data from the company's clinical trials for the purpose of legitimate scientific research. Requests for data may be addressed to datasharing@vaxcyte.com. Requests must be accompanied by a detailed analysis plan and will be reviewed for scientific validity. Data will be made available after initial product approval. Sharing of data may require execution of a data-sharing agreement.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be shared after deidentification and made available starting 6 months after initial product approval.
Access Criteria: Criteria will depend on the specific proposal received and may include qualification of the scientific researchers, potential contribution to the research field, scientific rigor of statistical and analytical methods, and other criteria appropriate for the proposal.